CLINICAL TRIAL: NCT02617251
Title: Impact of Deprivation on Hospital Care Efficiency in Paediatrics
Acronym: PRECAPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: PREPS -14-0530
Record Dates: First submitted 2015-11-19; First posted 2015-11-30 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2018-02

CONDITIONS: Deprivation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- neonatology patients: neonatology patients
  Interventions: Other: No intervention
- paediatric patients: paediatric patients
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Many studies have shown that deprived patients consumed more healthcare resources than non-deprived patients, in particular in terms of increased length of stay (LOS) and readmission rates, which has an impact on hospital efficiency and the healthcare system as a whole. There are many types of indicators available to assess deprivation in a hospital setting and French decision makers are currently using reliance on public aids to allocate additional funding to hospitals, based on the percentage of deprived patients they admit. However there are limits to this method: it only assesses one dimension of deprivation, the target population often does not know about the existence of those aids, and they have a clear threshold effect. An alternative solution is to use ecological deprivation indices which are obtained by aggregating different variables measured at a specific time and place, i.e. the patient's place of residence at the time of care. One such index, the FDep , was developed specifically in France, although others such as the Carstairs index and the European deprivation index also exist.

The primary objective of this study is to study the association between deprivation, measured by the FDep, and hospital care efficiency in paediatric and neonatology patients, measured by the difference between patient LOS and the national average LOS of their diagnosis-related group, DRG). The secondary objectives are to carry out a budget impact analysis on the impact of deprivation for hospitals with a paediatric or neonatology ward, to study the association between deprivation and readmission at 15 days, to study the relation between FDep and the currently used deprivation indicators, and to assess the added value of the FDep compared to those indicators and whether or not it should be used in routine practice.

In order to do so, an exhaustive retrospective study using the French hospital claims database will be carried out for the years 2012-2014. Deprivation indices will be calculated based on patients' postcode. The primary endpoint will be calculated using the national LOS present in the French national cost study. Similarly, the budget impact will look at the difference between production costs derived from the national cost study after adjusting for LOS and the statutory health insurance's tariffs, which will allow us to assess whether a hospital stay is associated with a gain, a loss or is budget-neutral for the hospital. Readmissions at 15 days will be identified through record linkage.

Descriptive analyses will summarise both hospital and patient characteristics. Uni- and bivariate analyses will be carried out by focusing of the variables of interest (e.g. average deprivation index by legal status of the hospital, mean LOS depending on the number of paediatric beds etc.). The deprivation index will be divided into quantiles as is the norm and the endpoints will be assessed for each of those quantiles. An ANOVA (or a Kruskal-Wallis test if the ANOVA hypotheses are not met) will test whether the results differ between each quantile. For readmission rates, a Chi² test will be performed.

In order to study the association between deprivation and the endpoints, the investigators will model each endpoint using as the main explanatory variable the deprivation index. Three main types of explanatory variables will be added to the model: patient characteristics (age, sex, severity level etc.), hospital characteristics (legal status, size, number of full-time equivalent etc.) and environment/context characteristics (number of paediatricians for 1,000 inhabitants, rural vs. urban area etc.).

In order to assess the added benefit of using the deprivation index vs. the current indicators, a sub-cohort will be constructed in Paris teaching hospitals (AP-HP) as unfortunately, whether the patient receives public aids is not present in the hospital claim database but is available only at the local level. The investigators will look at the distribution of patients with public aids in each quantile of the deprivation index and run the previous models using the two types of indicators one after the other and comparing the statistical performance of each pair of models.

ELIGIBILITY:
Inclusion Criteria:

Neonatology population

* Hospital stay present in the national hospital claims database in 2012-2014
* With a DRG and/or principal diagnosis related to neonatology
* In a hospital with a neonatology ward (including ICU)
* Age <28 days

Paediatric population

* Hospital stay present in the national hospital claim database in 2012-2014
* In a hospital with at least one paediatric department
* Age < 15 years old
* After exclusion of the neonatology stays previously identified

Exclusion Criteria:

* Day admissions
* Stays with error codes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospitalization in neonatology and pediatrics
Sampling Method: Non-Probability Sample
Enrollment: 3500000 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Hospital stay duration for participants | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Carel, MD-PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

REFERENCES:
- [Result] Michel M, Alberti C, Carel JC, Chevreul K. Association of Pediatric Inpatient Socioeconomic Status With Hospital Efficiency and Financial Balance. JAMA Netw Open. 2019 Oct 2;2(10):e1913656. doi: 10.1001/jamanetworkopen.2019.13656. PMID 31626320